CLINICAL TRIAL: NCT07018336
Title: Comparison of the Acute Effects of Mirror Therapy and Virtual Reality Therapy on Upper Extremity Function and Performance in Hemiplegic Patients
Brief Title: Mirror vs Virtual Reality Therapy for Upper Extremity Function in Hemiplegic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Çiçek Günday, Asst. Prof., Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07032025535
Record Dates: First submitted 2025-05-16; First posted 2025-06-12 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Hemiplegia; Stroke; Upper Extremity Dysfunction
Keywords: Stroke; Spasticity; Proprioception; Reaction Time
MeSH Terms: conditions — Hemiplegia; Stroke; Muscle Spasticity | interventions — Mirror Movement Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Other: Mirror Therapy
- Group B (Experimental)
  Interventions: Other: Virtual Reality (VR) Therapy

INTERVENTIONS:
Other: Mirror Therapy — Mirror Therapy will be applied to the affected upper extremity of hemiplegic patients by placing a mirror in the midsagittal plane, reflecting movements of the non-paretic limb to create the illusion that both limbs are moving symmetrically. Each session will include task-specific, functional hand and arm movements (e.g., grasping, wrist flexion/extension) performed for 30 minutes. Patients will be instructed to focus on the mirror image while actively engaging in the exercises.
  Arms: Group A
Other: Virtual Reality (VR) Therapy — Virtual Reality (VR) therapy will consist of a single 30-minute immersive session designed to engage the upper extremity of hemiplegic patients. Participants will wear a VR headset and interact with a virtual environment using motion-tracking controllers. Activities are task-oriented and aim to stimulate functional movement through simulated real-life scenarios (e.g., reaching, grabbing, stacking). This intervention offers multisensory feedback and high user engagement.
  Arms: Group B

SUMMARY:
Upper extremity impairment in hemiplegic patients significantly impacts daily activities and reduces quality of life. Although traditional rehabilitation methods can help, some patients experience limited progress. Recently, modern techniques such as mirror therapy and virtual reality (VR) have emerged, demonstrating promising results in motor skill improvement.

This study aims to directly compare the acute effects of mirror therapy and VR therapy on upper limb motor function in hemiplegic patients. Forty-two participants aged 18-75 with hemiplegia due to stroke (6-12 months post-stroke) will be randomly assigned to either mirror therapy or VR therapy. The evaluation includes motor function (Fugl-Meyer Assessment), spasticity (Modified Ashworth Scale), activities of daily living (Barthel Index), fine motor skills (Box and Block Test), proprioception, and reaction time.

The goal is to identify the effectiveness of the mirror therapy and VR therapy on motor function, spasticity control, proprioception, daily activity performance, and reaction times, contributing valuable insights to clinical rehabilitation practices.

DETAILED DESCRIPTION:
This study aims to comprehensively investigate and directly compare the immediate neurophysiological and functional effects of two innovative neurorehabilitation techniques-mirror therapy and virtual reality (VR) therapy-on upper extremity motor function among patients with hemiplegia following stroke. A total of 42 participants diagnosed with hemiplegia post-stroke will be randomly assigned to either Group A or Group B. Each participant will receive a single, structured intervention session lasting 30 minutes, designed to promote immediate motor recovery through targeted neuroplasticity-enhancing tasks.

Group A : Mirror Therapy Protocol: Participants will be seated comfortably in a stable and ergonomically supportive chair. A mirror measuring approximately 40 cm by 50 cm will be strategically positioned along the mid-sagittal plane, effectively reflecting the unaffected limb and creating the visual illusion of bilateral symmetrical movements. This visual feedback aims to activate motor-related cortical regions within the affected hemisphere, thus enhancing immediate functional motor improvements. Participants will engage in structured therapeutic exercises, each carefully designed to target various aspects of upper limb motor function:

* Reaching Task: Participants will perform reaching movements towards standardized objects positioned at varying distances and spatial orientations. They will complete 3 sets of 10 repetitions, progressively challenging their spatial accuracy, visual-motor integration, and motor planning skills.
* Joint Range Movements: Participants will execute comprehensive movements involving finger flexion-extension, wrist flexion-extension, elbow flexion-extension, and shoulder flexion-abduction. Each movement will be repeated 10 times, systematically activating multiple joints and muscles to promote functional range of motion and coordination.
* Grasp and Release Exercises: Participants will complete grasping and releasing tasks with objects of different sizes, textures, and weights. This task includes 3 sets of 10 repetitions designed to enhance tactile feedback, grip strength, fine motor coordination, and functional hand dexterity.

Group B: Virtual Reality (VR) Therapy: Participants in the VR group will utilize advanced virtual reality equipment, including high-resolution VR headsets and handheld controllers, immersing themselves in an interactive, three-dimensional virtual environment. This environment is specifically developed to simulate realistic and engaging scenarios, enhancing ecological validity, motivation, and patient engagement through multisensory stimulation. Therapeutic tasks in the VR environment will mirror those in the mirror therapy protocol to facilitate direct comparative analysis:

* Virtual Reaching Tasks: Participants will perform interactive tasks, engaging in accurate reaching movements toward virtual targets displayed at various locations and distances within the virtual environment, emphasizing hand-eye coordination and spatial orientation.
* Virtual Joint Movements: Virtual tasks will guide participants through movements involving finger flexion-extension, wrist flexion-extension, elbow flexion-extension, and shoulder flexion-abduction. Visual and auditory cues in the VR environment will enhance proprioceptive feedback and facilitate precise motor execution.
* Virtual Grasp and Release Tasks: Participants will virtually grasp and manipulate various digital objects, practicing controlled grasp and release movements that mimic real-world functional tasks. Task complexity will vary to address different aspects of motor control, strength, and dexterity.

Assessment Methods: Objective and reliable clinical assessments will be conducted immediately before and after each therapy session to measure changes in motor function, muscle tone, sensory-motor integration, and functional independence. The assessments will include:

* Motor Performance: Evaluated by the Fugl-Meyer Motor Assessment (FMA), providing comprehensive data on upper limb motor function.
* Spasticity: Quantified using the Modified Ashworth Scale (MAS), providing reliable measurements of muscle tone.
* Activities of Daily Living (ADL): Assessed with the Barthel Index to objectively measure functional independence and performance in daily activities.
* Fine Motor Skills: Evaluated using the Box and Block Test, offering precise measurement of hand dexterity and coordination.
* Proprioception: Evaluated using standardized joint position matching tasks, assessing sensory-motor integration and proprioceptive accuracy.
* Reaction Time: Assessed via computerized Simple Reaction Time (SRT) testing, precisely measuring sensorimotor responsiveness and processing speed.

This multidimensional assessment approach ensures a detailed evaluation of the acute therapeutic impacts of each intervention. By systematically comparing the immediate effectiveness and therapeutic advantages of mirror therapy and virtual reality therapy, this study aims to generate evidence-based recommendations, contributing significantly to clinical decision-making processes and potentially optimizing rehabilitation strategies for individuals recovering from stroke-related hemiplegia.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic patients in need of upper extremity rehabilitation.
* Having had a stroke 6 to 12 months prior to the study.
* Being at least Stage 3 for the upper extremity according to the Brunnstrom motor recovery stages.
* Age range: between 18 and 75 years.
* Individuals who volunteer to participate in the study.
* Individuals who are cognitively suitable for mirror therapy and virtual reality applications (a score of at least 24 on the Mini Mental State Examination)

Exclusion Criteria:

* Patients with severe spasticity (score ≥ 3 on the Modified Ashworth Scale)
* Individuals with secondary neurological conditions (e.g., Parkinson's disease, multiple sclerosis).
* Individuals diagnosed with vestibular dysfunction (as virtual reality equipment may cause issues like nausea or dizziness).
* Individuals with communication issues, such as hearing or vision loss.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment for Upper Extremity (FMA-UE) | Day 1
  The Fugl-Meyer Assessment is a standardized and widely used tool designed to evaluate motor function, balance, sensation, and joint functioning in individuals with post-stroke hemiplegia. In this study, only the upper extremity motor domain will be used, which includes evaluation of movement, coordination, and reflex action of the shoulder, elbow, forearm, wrist, and hand. The assessment is scored on a 3-point ordinal scale: 0 (cannot perform), 1 (performs partially), and 2 (performs fully), with a maximum score of 66 indicating better motor recovery. Participants are seated or lying in a comfortable position during the test, and each movement is explained and demonstrated. The researcher scores the quality and completion of each movement. The FMA-UE is a valid and reliable measure of motor function and is widely used in stroke rehabilitation research
Box and Block Test (BBT) | Day 1
  The Box and Block Test (BBT) is a standardized assessment of unilateral gross manual dexterity. Participants are instructed to transfer as many wooden blocks as possible from one compartment of a box to the other within 60 seconds using one hand. The number of successfully transferred blocks is recorded as the score. The test is widely recognized for its simplicity, reliability, and sensitivity in detecting changes in motor function, especially in post-stroke patients. In this study, the BBT will be used to evaluate changes in upper extremity motor performance and coordination immediately before and after the intervention session.

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | Day 1
  The Modified Ashworth Scale (MAS) is used to assess muscle spasticity by measuring resistance during passive soft-tissue stretching. It is a reliable clinical tool commonly used in neurological rehabilitation settings, especially in stroke patients. During the assessment, the target limb is passively moved through its range of motion, and the resistance to movement is rated on a 6-point scale ranging from 0 (no increase in muscle tone) to 4 (affected part rigid in flexion or extension). Participants are placed in a neutral and relaxed position during testing to ensure consistency. The evaluation will be conducted on the upper extremity muscles involved in voluntary function, and changes in MAS scores will be recorded to determine immediate effects of the intervention on spasticity levels.
joint Position Sense Test (Proprioception Assessment) | Day 1
  The Joint Position Sense Test assesses proprioceptive accuracy by evaluating a participant's ability to replicate specific joint angles with the opposite limb while blindfolded or with eyes closed. For this study, the test involves passive positioning of the affected upper limb at predetermined target angles (e.g., 60° and 100° of shoulder flexion), which participants will then attempt to match with the contralateral limb. The difference in angle reproduction is used as a measure of proprioceptive acuity. This method provides insight into sensorimotor integration deficits common in hemiplegic patients and will be used to assess changes before and after the intervention
Simple Reaction Time (SRT) with BlazePod | Day 1
  Simple Reaction Time (SRT) is a measure of how quickly an individual responds to a single stimulus. In this study, SRT will be evaluated using BlazePod light pods, which emit visual cues in a random sequence. Participants, seated comfortably with their hands resting near the pods, will be instructed to tap the lit pod as quickly as possible upon activation. The device records the reaction time in milliseconds. This test provides valuable information about the efficiency of sensorimotor integration and central processing speed. It is particularly relevant in stroke rehabilitation, where improvements in reaction time often correlate with better functional recovery.
Global Rating of Change (GRC) scale | Day 1
  The Global Rating of Change (GRC) scale is a subjective measure used to evaluate a patient's perceived improvement or deterioration in their health status over time. It is particularly useful in musculoskeletal and neurorehabilitation studies. In this study, participants will be asked to compare their current condition to their pre-treatment condition immediately after the therapy session. The version used includes a 5-point Likert scale ranging from -2 to +2, where: -2 = much worse, -1 = slightly worse, 0 = no change, +1 = slightly better, and +2 = much better. This simple, patient-centered outcome allows us to capture overall satisfaction and perceived effectiveness of the therapy from the patient's perspective.
Barthel Index (Activities of Daily Living - ADL) | Day 1
  The Barthel Index evaluates a patient's ability to perform basic activities of daily living (ADLs) independently. It assesses ten functional areas including feeding, bathing, grooming, dressing, bowel and bladder control, toilet use, transfers, mobility, and stair climbing. Each task is scored according to the level of assistance required, with a maximum total score of 100 indicating complete independence. The index is widely used in stroke rehabilitation to assess functional outcomes and monitor improvements over time. In this study, the Barthel Index will be administered before and immediately after the intervention to measure short-term functional changes in ADL performance among hemiplegic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Çiçek Günday, Asst. Prof., Principal Investigator — Istinye University, Department of Physiotherapy and Rehabilitation; Maysaa Hamdy Othman Ibrahim, Physiotherapist, Study Director — Istinye University, Department of Physiotherapy and Rehabilitation
Locations (1):
- İstinye Üniversite Hastanesi Medical Park Gaziosmanpaşa, Istanbul, Gaziosmanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No